CLINICAL TRIAL: NCT02346136
Title: Health Outcomes of Tai Chi in Subsidized Senior Housing
Acronym: Mi-WISH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: Brigham and Women's Hospital (Other); Brandeis University (Other); Massachusetts General Hospital (Other); University of Massachusetts, Boston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2R01AG025037-09A1 (NIH)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2018-04

CONDITIONS: Aging
Keywords: Tai Chi; Cluster randomized controlled trial; Intervention; Elderly; Mobility; Health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): This arm will receive a 6-month Tai Chi training intervention. Tai Chi training will include gentle dynamic stretching and strengthening, slow integrated movements, efficient posture, heightened body awareness and inner focus, active relaxation of body and mind, mindful diaphragmatic breathing, and healing imagery and intention. Participants will be asked to complete two formal group classes each week for at least 6 months, led by senior Tai Chi instructors. Additionally, participants will be given practice Digital Versatile Disc (DVD), DVD players if necessary, and instructions for daily home practice a minimum of 20 minutes on 3 non-class days each week.
  Interventions: Behavioral: Tai Chi training
- Educational Control (Active Comparator): This arm will receive a 6-month educational control intervention. Participants will attend monthly educational group sessions within a common area of each housing facility. Sessions will be led by research personnel and include material from Patient Education Forms (PEFs) produced by the American Geriatric Society. Sessions will be semi-structured and contain approximately 30 minutes of lecture and 30 minutes of group discussion.
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: Tai Chi training
  Arms: Tai Chi
Behavioral: Educational Control
  Arms: Educational Control

SUMMARY:
The proposed study will determine whether Tai Chi is an effective and practical intervention to improve overall function and lower health care utilization in an expensive, vulnerable population of seniors that is more representative of many US communities than those previously studied. If the results are favorable, our study will also provide the necessary training and protocol manuals to replicate Tai Chi programs in senior housing facilities across the nation to help prevent, better manage, and overcome frailty among seniors.

DETAILED DESCRIPTION:
Elderly people living in low-income housing facilities represent one of our nation's largest, most functionally impaired, economically disadvantaged, and understudied populations that account for a disproportionate share of Medicare spending. This trial aims to test whether Tai Chi exercises improve the health and reduce the health care utilization of this population more than health education and social calls by conducting a cluster randomized controlled trial in 16 housing facilities in cities surrounding Boston. The proposal builds upon previously successful studies by Drs. Lipsitz, Wayne, and others showing multiple benefits of Tai Chi exercises in elderly people with a variety of diseases and disabilities. A randomized, controlled pilot study showed that 12 weeks of Tai Chi exercises tailored to the abilities of frail seniors living in supportive housing facilities can improve balance, gait, and physical function. The proposed study aims are to determine the effects of Tai Chi exercises conducted at least twice weekly over a 6-month period on 1) functional performance measured by the Short Physical Performance Battery and 2) health care utilization determined from self-reported emergency room visits and hospitalizations in poor, multiethnic, elderly residents of low income housing facilities. Secondary outcomes will include person-centered measures such as physical function, cognition, psychological well-being, falls, and self-efficacy. We hypothesize that compared to the control intervention, Tai Chi will significantly improve physical function and reduce health care utilization. This study will prepare the necessary training and protocol manuals for widespread dissemination of Tai Chi programs in housing facilities across the nation. It will also provide estimates of potential Medicare cost savings that can be used to justify future health insurance payments for this intervention.

ELIGIBILITY:
Inclusion Criteria:

* able to understand instructions in English
* able to participate safely in Tai Chi exercises at least twice a week
* expected to remain in the facility for 1 year
* are fee-for-service Medicare Beneficiaries for the 3 study years
* Able to stand/walk independently, without the help of another person

Exclusion Criteria:

* enrolled in a Program of All-Inclusive Care for the Elderly (PACE), or a Special Needs Plan, since this would make it difficult to isolate the effects of Tai Chi on health care utilization.
* Practice of Tai Chi for >3 years over lifetime, or more than weekly in prior 6 months
* any unstable or terminal illness (e.g., unstable cardiovascular disease, active cancer, unstable chronic obstructive pulmonary disease (COPD), advanced dementia, psychosis)
* inability to maintain posture sitting or standing
* inability to hear, see, or understand Tai Chi instructions and assessment questions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Lipsitz, MD, Principal Investigator — Director, Marcus Institute for Aging Research, Hebrew SeniorLife; Peter Wayne, PhD, Principal Investigator — Research Director, Osher Center, Brigham and Women's Hospital
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

REFERENCES:
- [Background] Wayne PM, Gagnon MM, Macklin EA, Travison TG, Manor B, Lachman M, Thomas CP, Lipsitz LA. The Mind Body-Wellness in Supportive Housing (Mi-WiSH) study: Design and rationale of a cluster randomized controlled trial of Tai Chi in senior housing. Contemp Clin Trials. 2017 Sep;60:96-104. doi: 10.1016/j.cct.2017.07.005. Epub 2017 Jul 8. PMID 28694204
- [Result] Lipsitz LA, Macklin EA, Travison TG, Manor B, Gagnon P, Tsai T, Aizpurua II, Lo OY, Wayne PM. A Cluster Randomized Trial of Tai Chi vs Health Education in Subsidized Housing: The MI-WiSH Study. J Am Geriatr Soc. 2019 Sep;67(9):1812-1819. doi: 10.1111/jgs.15986. Epub 2019 May 22. PMID 31116883

RESULTS

PARTICIPANT FLOW:
Groups:
- Tai Chi: This arm will receive a 6-month Tai Chi training intervention. Tai Chi training will include gentle dynamic stretching and strengthening, slow integrated movements, efficient posture, heightened body awareness and inner focus, active relaxation of body and mind, mindful diaphragmatic breathing, and healing imagery and intention. Participants will be asked to complete two formal group classes each week for at least 6 months, led by senior Tai Chi instructors. Additionally, participants will be given practice Digital Versatile Disc (DVD), DVD players if necessary, and instructions for daily home practice a minimum of 20 minutes on 3 non-class days each week.
  Tai Chi training
- Educational Control: This arm will receive a 6-month educational control intervention. Participants will attend monthly educational group sessions within a common area of each housing facility. Sessions will be led by research personnel and include material from Patient Education Forms (PEFs) produced by the American Geriatric Society. Sessions will be semi-structured and contain approximately 30 minutes of lecture and 30 minutes of group discussion.
  Educational Control
Period: Overall Study
Arm/Group | Tai Chi | Educational Control
Started | 93 | 87
Completed | 71 | 64
Not Completed | 22 | 23
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Death | 1 | 0
Not completed — Study termination | 14 | 18

BASELINE CHARACTERISTICS:
Groups:
- Tai Chi: This arm will receive a 6-month Tai Chi training intervention. Tai Chi training will include gentle dynamic stretching and strengthening, slow integrated movements, efficient posture, heightened body awareness and inner focus, active relaxation of body and mind, mindful diaphragmatic breathing, and healing imagery and intention. Participants will be asked to complete two formal group classes each week for at least 6 months, led by senior Tai Chi instructors. Additionally, participants will be given practice DVDs (and DVD players if necessary) and instructions for daily home practice a minimum of 20 minutes on 3 non-class days each week.
  Tai Chi training
- Total: Total of all reporting groups
Arm/Group | Tai Chi | Educational Control | Total
Number analyzed (Participants) | 93 | 87 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 14 | 23
  >=65 years | 84 | 73 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (9.1) | 74.6 (8.6) | 75.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 57 | 120
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 88 | 84 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 23 | 58
  White | 50 | 62 | 112
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 87 | 180
Short Physical Performance Battery Total Score [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery includes measures of standing balance (timing of tandem, semi-tandem, and side-by-side stands), 4-meter walking speed and the ability and time to rise from a chair 5 times. The minimum score = 0, the maximum score=12. A higher score means a better outcome.
  units on a scale | 7.92 (2.76) | 8.36 (2.89) | 8.14 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Physical Performance Battery (SPPB) Total Score
Description: The Short Physical Performance Battery includes measures of standing balance (timing of tandem, semi-tandem, and side-by-side stands), 4-meter walking speed and the ability and time to rise from a chair 5 times. The minimum score = 0, the maximum score=12. A higher score means a better outcome.
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
units on a scale | 0.05 (0.18) | 0.18 (0.19)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.62, Mixed Models Analysis — Tested as two-tailed p<0.025 to accommodate two co-primary outcomes; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.62 to 0.37], Standard Error of Mean 0.25

2. Primary Outcome: Health Care Utilization
Description: Health care utilization will be defined by counts of hospitalizations during the study period.
Time Frame: up to 12 months
Population: The 142 participants analyzed for health care utilization measures were those enrolled at sites that initiated assigned treatment (excluding 32 participants), had not withdrawn prior to treatment initiation (excludes 4 participants), and for whom at least one assessment of health care utilization was completed (excludes 2 participants).
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 75 | 67
Participants
  0 hospitalizations | 66 | 56
  1 hospitalization | 5 | 9
  2 hospitalizations | 2 | 2
  3 hospitalizations | 2 | 0
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.194, Mixed Models Analysis; Mixed model Poisson reg with fixed effects of age, baseline SPPB, baseline CES-D, and falls in prev year and random intercept and trt by site pair; Risk Ratio (RR) = 0.535, 95% CI 2-sided [0.182 to 1.57] — Numerator of risk ratio is the rate among participants at sites receiving Tai Chi. Denominator of risk ratio is the rate among participants at sites receiving Health Education

3. Secondary Outcome: Mobility
Description: Mobility will be assessed by the Timed Up-and-Go, which records the time needed to stand from a chair, walk three meters, turn, walk back to the chair and sit down.
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
seconds | .18 (.73) | .83 (.77)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = .50, Mixed Models Analysis; Mean Difference (Net) = -.65, 95% CI 2-sided [-2.53 to 1.24], Standard Error of Mean .94

4. Secondary Outcome: Gait Velocity
Description: Gait velocity will be measured in meters/second (m/s) during two conditions: Normal walking (NW) and Dual task(DT) condition (counting backwards by 3's or 1's while walking)
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
m/s
  Gait NW velocity | .01 (.02) | .01 (.02)
  Gait DT velocity | .02 (.01) | -.00 (.01)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Gait NW velocity variable; Test type: Superiority; p = .85, Mixed Models Analysis; Mean Difference (Net) = .00, 95% CI 2-sided [-.04 to .05], Standard Error of Mean .02
Statistical Analysis 2: Comparison: Tai Chi vs Educational Control; Gait DT velocity variable; Test type: Superiority; p = .26, Mixed Models Analysis; Mean Difference (Net) = .02, 95% CI 2-sided [-.02 to .06], Standard Error of Mean .02

5. Secondary Outcome: Standing Balance
Description: Standing balance will be assessed by recording 95% ellipse sway area with eyes open in meters squared (m2)
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: m^2
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
m^2 | 0.01 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = -0.004, 95% CI 2-sided [-0.04 to 0.03], Standard Error of Mean 0.02

6. Secondary Outcome: Grip Strength
Description: Grip strength of the dominant hand will be assessed with a hand-grip dynamometer in kilograms (kg).
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
kg | 0.64 (0.50) | -0.17 (0.52)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = .26, Mixed Models Analysis; Mean Difference (Net) = 0.81, 95% CI 2-sided [-0.61 to 2.22], Standard Error of Mean 0.71

7. Secondary Outcome: Self-reported Physical Activity
Description: Self-reported physical activity will be assessed with the Physical Activity Scale for the Elderly (PASE). The range for this scale is 0-400, with higher score representing higher activity score (better outcome).
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
scores on a scale | -3.42 (5.17) | -4.14 (5.37)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = .92, Mixed Models Analysis; Median Difference (Net) = .72, 95% CI 2-sided [-13.9 to 15.3], Standard Error of Mean 7.29

8. Secondary Outcome: Executive Function
Description: Executive function will be assessed with the Trail Making Test (TMT). Participants are timed while sequentially connecting a series of numbered circles (TMT part A), as well as connecting an alternating series of numbers and letters (e.g., A-1-B-2-C-3…) (TMT part B).
  The outcome measure is the time difference in seconds between Part B and Part A.
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
seconds | -8.19 (6.91) | -9.55 (7.37)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = .88, Mixed Models Analysis; Median Difference (Net) = 1.36, 95% CI 2-sided [-17.2 to 19.9], Standard Error of Mean 9.28

9. Secondary Outcome: Health-related Quality-of-life
Description: Health-related quality-of-life will be assessed with the Short Form-12 (SF-12), which is a 12 item short form survey, a shortened version of the Short Form-36 (SF-36) health survey that is widely-utilized to assess physical and mental health, as well as the outcomes of healthcare services. The total score ranges from 0-100, with a lower score representing a better outcome for *both* the "Physical component" and "Mental Component"
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
scores on a scale
  Physical component | .22 (.99) | -.64 (1.04)
  Mental component | -1.81 (1.16) | -.71 (1.19)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Physical component score; Test type: Superiority; p = .55, Mixed Models Analysis; Mean Difference (Net) = .85, 95% CI 2-sided [-2.00 to 3.71], Standard Error of Mean 1.43
Statistical Analysis 2: Comparison: Tai Chi vs Educational Control; Mental component score; Test type: Superiority; p = .51, Mixed Models Analysis; Mean Difference (Net) = -1.10, 95% CI 2-sided [-4.41 to 2.21], Standard Error of Mean 1.66

10. Secondary Outcome: Depression
Description: Depressive symptoms will be assessed with the Center of Epidemiology Studies-Depression Scale Revised (CESD-R). The 20 item CESD-R test score range is between 0-60, with a lower score representing a better outcome.
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
score on a scale | -.06 (.69) | -.47 (.74)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = .69, Mixed Models Analysis; Median Difference (Net) = .40, 95% CI 2-sided [-1.60 to 2.41], Standard Error of Mean 1.00

11. Secondary Outcome: Exercise Self-efficacy
Description: Exercise self-efficacy will be assessed with a valid and reliable exercise self-efficacy questionnaire (Activities-specific Balance Confidence (ABC) score). The ABC score ranges from 0-100, with a higher score indicating a better outcome.
Time Frame: Change from baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
score on a scale | 0.11 (1.77) | -2.02 (1.87)
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.41, Mixed Models Analysis — to accommodate two co-primary outcomes; Mean Difference (Net) = 2.14, 95% CI 2-sided [-2.98 to 7.26], Standard Error of Mean 2.56

12. Secondary Outcome: Falls
Description: Falls will be defined as any event in which the participant unintentionally comes to rest on the ground or other lower level, not as a result of a major intrinsic event or an overwhelmingly external hazard. This outcome measure is reporting the sum total number of falls for each intervention.
Time Frame: 12 months
Measure: Number; unit: falls
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 77 | 67
falls | 26 | 16

13. Secondary Outcome: Health Care Utilization
Description: Secondary health care utilization outcomes include counts of emergency room visits.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 75 | 67
Participants
  0 ED visits | 55 | 45
  1 ED visit | 15 | 10
  2 ED visits | 4 | 8
  3 ED visits | 0 | 3
  5 ED visits | 1 | 0
  8 ED visits | 0 | 1
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.060, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.476, 95% CI 2-sided [0.216 to 1.05] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Mini-Mental State Examination
Description: The Mini-Mental State Questionnaire is a 30 point questionnaire that is used extensively to measure cognitive impairment. Total score = 30, score ranges are from 0 to 30. A higher score indicates better performance.
Time Frame: Change from baseline to 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tai Chi | Educational Control
Number analyzed (Participants) | 93 | 87
score on a scale | 0.89 [-0.34 to 2.11] | -0.38 [-1.58 to 0.82]
Statistical Analysis 1: Comparison: Tai Chi vs Educational Control; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = 1.27, 95% CI 2-sided [-0.40 to 2.94], Standard Error of Mean 0.81

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 1 year
Arm/Group | Tai Chi | Educational Control
All-Cause Mortality (participants affected / at risk) | 3/77 | 0/67
Serious Adverse Events (participants affected / at risk) | 13/77 | 8/67
Other Adverse Events (participants affected / at risk) | 44/77 | 12/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi (N=77) | Educational Control (N=67)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi (N=77) | Educational Control (N=67)
Fall (Injury, poisoning and procedural complications) | 21 (26) | 11 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 18 (21) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT02346136/Prot_SAP_000.pdf